CLINICAL TRIAL: NCT02160145
Title: A Phase 3b, Multi-center, Randomized-withdrawal, Placebo-controlled, Double-blind, Parallel-group Trial to Compare the Efficacy and Safety of Tolvaptan (45 to 120 mg/Day, Split-dose) in Subjects With Chronic Kidney Disease Between Late Stage 2 to Early Stage 4 Due to Autosomal Dominant Polycystic Kidney Disease
Brief Title: Efficacy and Safety of Tolvaptan in Subjects With Chronic Kidney Disease Between Late Stage 2 to Early Stage 4 Due to Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-13-210
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Chronic Kidney Disease; Autosomal Dominant Polycystic Kidney Disease
Keywords: Chronic Kidney Disease; Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan (Experimental): Tolvaptan (OPC-41061)
  Interventions: Drug: Tolvaptan (OPC-41061)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan (OPC-41061) — Tolvaptan tablets (15 or 30 mg) will be self-administered orally as split-dose regimens, once upon awakening and another approximately 8 to 9 hours later.
  Arms: Tolvaptan
Drug: Placebo — Matching placebo tablets will be self-administered orally as split-dose regimens, once upon awakening and another approximately 8 to 9 hours later
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether tolvaptan is effective and safe for the treatment of late-stage chronic kidney disease due to autosomal dominant polycystic kidney disease (ADPKD)

DETAILED DESCRIPTION:
The protocol will extend the understanding of the efficacy and safety of tolvaptan treatment in ADPKD patients with late stage 2 to early stage 4 CKD (chronic kidney disease).

This trial will compare the efficacy of tolvaptan treatment in reducing the annualized change in estimated glomerular filtration rate (eGFR) from pre-treatment baseline to post-treatment follow-up, as compared with placebo, in subjects who tolerate tolvaptan during an initial run-in period. The change in eGFR, calculated by the Chronic Kidney Disease-Epidemiology (CKD-EPI) formula, will provide kidney function data that are complementary to the data demonstrating the benefits previously observed primarily in ADPKD subjects with earlier stages of disease.

Also, it will compare the efficacy of tolvaptan treatment in reducing the decline of annualized eGFR slope, as compared with placebo, in this type of subjects. Finally, it will compare the overall and hepatic safety profile of tolvaptan with placebo and to compare incidence of ADPKD complications (outcomes) during the trial

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with eGFR between 25-65 mL/min/1.73m2 (if aged 18 to55) or eGFR between 25-44 mL/min/1.73m2 (if aged 56 to <66)
* Tolvaptan naïve
* Diagnosis of ADPKD by modified pei-Ravine criteria 1) 3 cysts per kidney by sonography or 5 cysts by CT or MRI with family history of ADPKD or 2) 10 cysts per kidney by any radiologic method and exclusion of other cystic kidney diseases if without family history

Exclusion Criteria:

* Women of childbearing potential who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days after the last dose of Investigational medicinal product (IMP)
* Women who are breast-feeding and/or who have a positive pregnancy test prior to receiving IMP
* Need for chronic diuretic use
* Hepatic impairment or liver function abnormalities other than that expected for ADPKD with typical cystic liver disease
* Advanced diabetes, evidence of additional significant renal disease, renal cancer, single kidney, recent renal surgery or acute kidney injury
* Contraindications to required trial assessments
* Medical history or medical findings inconsistent with safety or compliance with trial assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1370 (Actual)
Dates: Start 2014-05; Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (206):
- United States (76):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Denver, Colorado
  - New Haven, Connecticut
  - Hudson, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Ocala, Florida
  - Port Charlotte, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Meridian, Idaho
  - Chicago, Illinois
  - Kansas City, Kansas
  - Wichita, Kansas
  - Baton Rouge, Louisiana
  - Lafayette, Louisiana
  - Baltimore, Maryland
  - Greenbelt, Maryland
  - Rockville, Maryland
  - Wheaton, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Pontiac, Michigan
  - Roseville, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Reno, Nevada
  - Eatontown, New Jersey
  - Voorhees Township, New Jersey
  - Buffalo, New York
  - Mineola, New York
  - New York, New York
  - Rosedale, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Grand Forks, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Bethlehem, Pennsylvania
  - Doylestown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Orangeburg, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - McAllen, Texas
  - Burlington, Vermont
  - Arlington, Virginia
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Wenatchee, Washington
  - Morgantown, West Virginia
  - La Crosse, Wisconsin
- Argentina (7):
  - Bahía Blanca, Buenos Aires
  - Ciudad Autonoma, Buenos Aires
  - Junín, Buenos Aires
  - Pergamino, Buenos Aires
  - Pilar, Buenos Aires
  - Sarandí, Buenos Aires
  - Córdoba
- Australia (12):
  - Camperdown, New South Wales
  - Concord, New South Wales
  - New Lambton Heights, New South Wales
  - St Leonards, New South Wales
  - Westmead, New South Wales
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Launceston, Tasmania
  - Parkville, Victoria
  - Reservoir, Victoria
  - Richmond, Victoria
  - Perth, Western Australia
- Belgium (7):
  - Aalst
  - Antwerp
  - Brussels
  - Ghent
  - Kortrijk
  - Leuven
  - Liège
- Canada (6):
  - Edmonton, Alberta
  - St. John's, Newfoundland and Labrador
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
- Czechia (9):
  - Brno
  - České Budějovice
  - Hradec Králové
  - Jihlava
  - Jilemnice
  - Liberec
  - Ostrava
  - Prague
  - Tábor
- Denmark (5):
  - Aalborg
  - Aarhus C
  - Holstebro
  - Odense C
  - Viborg
- France (10):
  - Brest, Finistere
  - Bordeaux, Gironde
  - Toulouse, Haute Garonne
  - Montpellier, Herault
  - Grenoble, Isere
  - Reims, Marne
  - Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Saint-Priest-En-Jarez, Pays de la Loire Region
  - Lyon, Rhone
  - Pierre-Bénite, Rhone
- Germany (8):
  - Heidelberg, Baden-Wurttemberg
  - Munich, Bavaria
  - Nuremberg, Bavaria
  - Hanover, Lower Saxony
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Wiesbaden, North Rhine-Westphalia
  - Dresden, Saxony
- Hungary (3):
  - Budapest
  - Pécs
  - Szeged
- Israel (6):
  - Ashkelon
  - Jerusalem
  - Nahariya
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (9):
  - Torrette Di Ancona, Ancona
  - Montichiari, Brescia
  - Bari
  - Bologna
  - Lecco
  - Milan
  - Modena
  - Napoli
  - Pavia
- Netherlands (2):
  - Groningen
  - Nijmegen
- Norway (3):
  - Bergen
  - Oslo
  - Stavanger
- Poland (7):
  - Ciechanów
  - Golub-Dobrzyń
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
  - Wroclaw
- San Juan, Puerto Rico
- Romania (2):
  - Bucharest
  - Oradea
- Russia (3):
  - Krasnoyarsk
  - Saint Petersburg
  - Yaroslavl
- South Africa (3):
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
- Spain (5):
  - L'Hospitalet de Llobregat, Barcelona
  - Ciudad Real
  - Madrid
  - Seville
  - Valencia
- Sweden (5):
  - Gothenburg
  - Linköping
  - Örebro
  - Stockholm
  - Uppsala
- United Kingdom (17):
  - Exeter, Devon
  - Hull, East Riding Of Yorkshire
  - Brighton, East Sussex
  - London, Greater London
  - Manchester, Greater Manchester
  - Salford, Greater Manchester
  - Stevenage, Hertfordshire
  - Inverness, Highland Region
  - Leicester, Leicestershire
  - Edinburgh, Lothian Region
  - Liverpool, Merseyside
  - Middlesbrough, North Yorkshire
  - Sheffield, South Yorkshire
  - Stoke-on-Trent, Staffordshire
  - Newcastle upon Tyne, Tyne & Wear
  - Coventry, Warwickshire
  - Swansea

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Chebib FT, Zhou X, Garbinsky D, Davenport E, Nunna S, Oberdhan D, Fernandes A. Tolvaptan and Kidney Function Decline in Older Individuals With Autosomal Dominant Polycystic Kidney Disease: A Pooled Analysis of Randomized Clinical Trials and Observational Studies. Kidney Med. 2023 Apr 14;5(6):100639. doi: 10.1016/j.xkme.2023.100639. eCollection 2023 Jun. PMID 37250503
- [Derived] Alpers DH, Lewis JH, Hunt CM, Freston JW, Torres VE, Li H, Wang W, Hoke ME, Roth SE, Westcott-Baker L, Estilo A. Clinical Pattern of Tolvaptan-Associated Liver Injury in Trial Participants With Autosomal Dominant Polycystic Kidney Disease (ADPKD): An Analysis of Pivotal Clinical Trials. Am J Kidney Dis. 2023 Mar;81(3):281-293.e1. doi: 10.1053/j.ajkd.2022.08.012. Epub 2022 Sep 30. PMID 36191725
- [Derived] Bennett H, McEwan P, Hamilton K, O'Reilly K. Modelling the long-term benefits of tolvaptan therapy on renal function decline in autosomal dominant polycystic kidney disease: an exploratory analysis using the ADPKD outcomes model. BMC Nephrol. 2019 Apr 23;20(1):136. doi: 10.1186/s12882-019-1290-5. PMID 31014270
- [Derived] Torres VE, Chapman AB, Devuyst O, Gansevoort RT, Perrone RD, Koch G, Ouyang J, McQuade RD, Blais JD, Czerwiec FS, Sergeyeva O; REPRISE Trial Investigators. Tolvaptan in Later-Stage Autosomal Dominant Polycystic Kidney Disease. N Engl J Med. 2017 Nov 16;377(20):1930-1942. doi: 10.1056/NEJMoa1710030. Epub 2017 Nov 4. PMID 29105594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject first visit: 21 May 2014; Last subject last visit: 18 April 2017. Subjects were recruited from 213 sites in 21 countries. Of 2292 subjects screened, 1519 entered the 6-week run-in period; 23 were placebo run-in failures and 126 were tolvaptan titration/run-in failures.
Pre-assignment Details: Subjects with Stage 2 - 4 chronic kidney disease (CKD) due to Autosomal Dominant Polycystic Kidney Disease (ADPKD) were stratified by baseline estimated glomerular filtration rate (eGFR) (≤ 45 or > 45 milliliters/minute/ 1.73 square metres [mL/min/1.73 m^2]), by age (≤ 55 or > 55 years), and total kidney volume (≤ 2000 mL, > 2000 mL, or unknown).
Groups:
- All Subjects Prerandomization: Following screening, the single-blind prerandomization period (Day -42 to Day -1) consisted of:
  1. Placebo Run-in: All subjects received a daily split-dose of placebo (0/0 milligrams [mg]) in a form identical to 15/15 mg tolvaptan split-dose for 1 week.
  2. Tolvaptan Titration: Over 2 weeks all subjects received a split-dose of 30/15 mg (2 x 15mg tablets upon waking, then 1 x 15 mg tablet 8-9 hours later) which was titrated up every 3-4 days to 45/15 mg, then 60/30 mg, and up to a maximum dose of 90/30 mg.
  3. Tolvaptan Run-in: Eligible subjects who tolerated at least 60/30 mg tolvaptan during titration entered the 3-week run-in period and continued on a stable dose of 60/30 mg or 90/30 mg tolvaptan to confirm eligibility and establish prerandomization baseline.
- Tolvaptan: Double-blind Randomized Treatment Period (Day 0 to Month 12): Following randomization subjects continued on the same dose of tolvaptan they received during the tolvaptan run-in period (60/30 mg or 90/30 mg) for a duration of 12 months.
  Follow-up Period: A 3-week final follow-up for efficacy analysis.
- Placebo: Double-blind Randomized Treatment Period (Day 0 to Month 12):
  Following randomization subjects received placebo tablets matching their tolerated tolvaptan dose during the tolvaptan run-in period (60/30 mg or 90/30 mg) for a duration of 12 months.
  Follow-up Period: A 3-week final follow-up for efficacy analysis.
Period: Prerandomization Single-blind Period
Arm/Group | All Subjects Prerandomization | Tolvaptan | Placebo
Started | 1519 | 0 | 0
Treated in Placebo Run-in | 1514 | 0 | 0
Treated in Tolvaptan Titration/Run-in | 1491 | 0 | 0
Randomized | 1370 | 0 | 0
Completed | 1370 | 0 | 0
Not Completed | 149 | 0 | 0
Not completed — Placebo run-in failure | 23 | 0 | 0
Not completed — Tolvaptan titration/run-in failure | 126 | 0 | 0
Period: Randomized Double-blind Period
Arm/Group | All Subjects Prerandomization | Tolvaptan | Placebo
Started | 0 (1370 subjects were randomized to receive tolvaptan or placebo in the double-blind period.) | 683 (Subjects completed the single-blind period and were randomized to receive tolvaptan.) | 687 (Subjects completed the single-blind period and were randomized to receive placebo.)
On-treatment Completers | 0 | 578 | 637
Off-treatment Completers | 0 | 76 | 22
Completed (Completed Month 12 Visit) | 0 | 654 | 659
Not Completed | 0 | 29 | 28
Not completed — Subject decision | 0 | 21 | 20
Not completed — Lost to Follow-up | 0 | 1 | 3
Not completed — Physician Decision | 0 | 7 | 5

BASELINE CHARACTERISTICS:
Population: The baseline population consisted of all randomized subjects.
Arm/Group | Tolvaptan | Placebo | Total Title
Number analyzed (Participants) | 683 | 687 | 1370
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (8.2) | 47.2 (8.2) | 47.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 336 | 354 | 690
  Male | 347 | 333 | 680
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 35 | 79
  Not Hispanic or Latino | 632 | 647 | 1279
  Unknown or Not Reported | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 22 | 19 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 23 | 48
  White | 626 | 632 | 1258
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: The Mean Annualized Change in eGFR From Pretreatment Baseline to Post-treatment Follow-up.
Description: The mean annualized change in eGFR was calculated using the Chronic Kidney Disease-Epidemiology (CKD-EPI) formula from pretreatment baseline to post-treatment follow-up, annualized (divided) by each subject's trial duration.
  The baseline for the primary endpoint was defined as the average of up to 3 eGFR values observed during the screening and placebo run-in periods.
Time Frame: Pretreatment baseline to post-treatment follow-up (up to 61 weeks).
Population: The primary endpoint efficacy population consisted of all subjects who were in the randomized sample, took at least 1 dose of investigational medicinal product (IMP) after randomization, and had a baseline and at least 1 valid post-treatment evaluation in eGFR (i.e at least 1 week off-treatment).
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2/year
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 668 | 663
mL/min/1.73 m^2/year | -2.339 (0.240) | -3.610 (0.240)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Tolvaptan versus placebo. Treatment difference in the change of eGFR assessed the efficacy of tolvaptan treatment as compared with placebo in subjects with late-stage CKD due to ADPKD who tolerated tolvaptan during an initial run-in period; Test type: Other; p < 0.0001, ANCOVA — A 2-sided alpha of 0.05 was applied to the primary analysis of the primary endpoint; Weighted Analysis of Covariance (ANCOVA) with effects of treatment and randomization stratification factors and covariate baseline; Treatment difference = 1.271, 95% CI 2-sided [0.859 to 1.684]

2. Secondary Outcome: Mean Annualized Slope of eGFR Change
Description: To compare the efficacy of tolvaptan treatment in reducing the decline of annualized eGFR slope, as compared with placebo, in subjects with late-stage CKD due to ADPKD who tolerated tolvaptan during an initial run-in period, the annualized rate of eGFR change was derived from each individual subject's eGFR slope using the CKD-EPI formula.
  The annualized eGFR change slope was derived from all eGFR observations from placebo-run-in, tolvaptan run-in, double-blind treatment and post-treatment follow-up periods using the linear mixed model of analysis. The mean annualized slope of eGFR change is presented.
Time Frame: Pretreatment baseline to post-treatment follow-up (up to 61 weeks).
Population: The key secondary endpoint efficacy population consisted of all randomized subjects who took at least 1 dose of IMP after randomization, and have a baseline (average of up to 3 eGFR values observed during screening and placebo run-in periods) and at least 1 post-randomization evaluation in eGFR during the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2/year
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 680 | 682
mL/min/1.73m^2/year | -3.160 (0.140) | -4.170 (0.142)
Statistical Analysis 1: Comparison: Tolvaptan vs Placebo; Difference in treatment effect was derived from a linear mixed model with effects of treatment, time, treatment ime interaction, acute haemodynamic effect, pretreatment baseline, and randomization stratification factors. An unstructured variance matrix was assumed for the random intercept and time; Test type: Other; p < 0.0001, Mixed Models Analysis — A two-sided alpha of 0.05 was applied when the primary endpoint reached a two-sided alpha of 0.05; Treatment difference = 1.011, 95% CI 2-sided [0.618 to 1.403]

3. Other Pre Specified Outcome: Mean Change From Baseline in Urine Osmolality During the Double-blind Treatment Period and Post-treatment Follow-up
Description: The mean change from baseline in urine osmolality for the double-blind treatment period collection timepoints and post-treatment follow-up are presented. Baseline was defined as the last evaluation prior to post-randomization dosing.
Time Frame: Baseline and Months 3, 6, 9 and 12 (End of treatment visit) of the double-blind treatment period, and post-treatment follow-up.
Population: The primary safety population consisted of all subjects who were randomized and took at least 1 dose of IMP after randomization. Only subjects with data available for analysis at the timepoints of testing are presented.
Measure: Mean (Standard Deviation); unit: milliosmole per kilogram (mOSm/kg)
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 681 | 685
milliosmole per kilogram (mOSm/kg)
  Month 3: number analyzed (Participants) | 655 | 664
  Month 3 | 10.2 (80.3) | 177.7 (124.5)
  Month 6: number analyzed (Participants) | 637 | 652
  Month 6 | 22.9 (84.3) | 179.1 (126.2)
  Month 9: number analyzed (Participants) | 625 | 646
  Month 9 | 30.4 (92.1) | 179.9 (125.1)
  Month12: number analyzed (Participants) | 629 | 651
  Month12 | 36.9 (96.0) | 180.3 (121.1)
  Follow-up: number analyzed (Participants) | 624 | 650
  Follow-up | 162.4 (114.0) | 179.5 (128.9)

4. Other Pre Specified Outcome: Mean Change From Baseline in Urine Specific Gravity During the Double-blind Treatment Period and Post-treatment Follow-up
Description: The mean change from baseline in urine specific gravity for the double-blind treatment period collection timepoints and post-treatment follow up are presented. Baseline was defined as the last evaluation prior to post-randomization dosing.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 681 | 685
unitless
  Month 3: number analyzed (Participants) | 654 | 662
  Month 3 | 0.0001 (0.0022) | 0.0041 (0.0033)
  Month 6: number analyzed (Participants) | 638 | 649
  Month 6 | 0.0003 (0.0024) | 0.0042 (0.0033)
  Month 9: number analyzed (Participants) | 623 | 641
  Month 9 | 0.004 (0.0025) | 0.0040 (0.0032)
  Month 12: number analyzed (Participants) | 635 | 648
  Month 12 | 0.0006 (0.0027) | 0.0040 (0.0033)
  Follow-up: number analyzed (Participants) | 620 | 653
  Follow-up | 0.0037 (0.0031) | 0.0040 (0.0034)

ADVERSE EVENTS:
Time Frame: For the tolvaptan single-blind period: 35 days (Day -35 to Day -1). For the double-blind treatment period: 12 months (Day 0 to 12 months).
Description: Treatment emergent adverse events (AEs) were collected, defined as an AE that started after IMP treatment or an AE that was continuous from baseline and was serious, IMP related or resulted in death, discontinuation, interruption or reduction of IMP treatment.
Groups:
- Tolvaptan (Single-blind Treatment Period): The secondary safety population consisted of all subjects who took at least one dose of tolvaptan during the tolvaptan titration/run-in periods.
- Tolvaptan (Double-blind Treatment Period): The tolvaptan primary safety population consisted of all subjects who were randomized in the double-blind treatment period and who took at least one dose of tolvaptan after randomization.
- Placebo (Double-blind Treatment Period): The placebo primary safety population consisted of all subjects who were randomized in the double-blind treatment period and who took at least one dose of placebo after randomization.
Arm/Group | Tolvaptan (Single-blind Treatment Period) | Tolvaptan (Double-blind Treatment Period) | Placebo (Double-blind Treatment Period)
All-Cause Mortality (participants affected / at risk) | 1/1491 | 0/681 | 1/685
Serious Adverse Events (participants affected / at risk) | 43/1491 | 85/681 | 60/685
Other Adverse Events (participants affected / at risk) | 1051/1491 | 581/681 | 564/685
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolvaptan (Single-blind Treatment Period) (N=1491) | Tolvaptan (Double-blind Treatment Period) (N=681) | Placebo (Double-blind Treatment Period) (N=685)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Congenital Hepatic Fibrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Incarcerated Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Thirst (General disorders) | 2 (2) | 0 (0) | 0 (0)
Cyst rupture (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
HIV infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal cyst infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (4) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Hepatic cyst infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 8 (8) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Liver function test abnormal (Investigations) | 1 (1) | 3 (3) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 11 (12) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 4 (7) | 2 (2)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral artery thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Nocturia (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 2 (2) | 3 (3) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3)
Renal pain (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (3)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolvaptan (Single-blind Treatment Period) (N=1491) | Tolvaptan (Double-blind Treatment Period) (N=681) | Placebo (Double-blind Treatment Period) (N=685)
Dry mouth (Gastrointestinal disorders) | 132 (134) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 47 (54) | 23 (25)
Thirst (General disorders) | 430 (453) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 46 (49) | 24 (27)
Oedema peripheral (General disorders) | 0 (0) | 30 (37) | 45 (50)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 59 (70) | 58 (71)
Urinary tract infection (Infections and infestations) | 0 (0) | 39 (48) | 55 (65)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 72 (98) | 84 (111)
Blood creatinine increased (Investigations) | 0 (0) | 46 (58) | 46 (56)
Polydipsia (Metabolism and nutrition disorders) | 146 (147) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 34 (37) | 41 (46)
Headache (Nervous system disorders) | 0 (0) | 55 (66) | 59 (65)
Nocturia (Renal and urinary disorders) | 308 (319) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 475 (488) | 36 (38) | 11 (11)
Haematuria (Renal and urinary disorders) | 0 (0) | 37 (52) | 35 (42)
Renal pain (Renal and urinary disorders) | 0 (0) | 113 (158) | 130 (174)
Hypertension (Vascular disorders) | 0 (0) | 73 (88) | 79 (96)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT02160145/SAP_000.pdf
  • Study Protocol (2015-03-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT02160145/Prot_001.pdf